CLINICAL TRIAL: NCT03294291
Title: Quadratus Lumborum Block Versus Caudal Block
Brief Title: Ultrasound Guided Quadratus Lumborum Block Versus Caudal Block in Pediatric Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Gözen Öksüz, Assistant Professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017/10-08
Record Dates: First submitted 2017-09-22; First posted 2017-09-27 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: All Children will be randomly assigned to one of 2 groups of 25 patients each using a computer-generated number table.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadratus Lumborum block group (Active Comparator): After preoxygenation for three minutes, anesthesia would be induced with 8% sevoflurane inhalation in 50% oxygen and % 50 air ; 1ug/kg fentanyl and 3 mg/kg propofol is administered intravenously. Then laryngeal mask is inserted when conditions are satisfactory. Under ultrasound guidance a 22 Gauge, Pajunk Sonoplex(medical Germany) needle will be used for both techniques. Under ultrasound 0.7 ml/kg bupivacaine 0.25 % injected unilaterally at the posterior border of the quadratus lumborum muscle.
  Interventions: Procedure: Quadratus lumborum block
- Caudal block (Active Comparator): After preoxygenation for three minutes, anesthesia would be induced with 8% sevoflurane inhalation in 50% oxygen and % 50 air ; 1ug/kg fentanyl and 3 mg/kg propofol is administered intravenously. Then laryngeal mask is inserted when conditions are satisfactory caudal block wil performe with bupivacaine 0.7 ml/kg as 0.25%.
  Interventions: Procedure: Caudal block

INTERVENTIONS:
Procedure: Quadratus lumborum block — Postoperative pain procedure
  Arms: Quadratus Lumborum block group
Procedure: Caudal block — Postoperative pain procedure
  Arms: Caudal block

SUMMARY:
The purpose of this research study is to find the best way to decrease pain in children whom have had low abdominal surgery. Investigators will perform two technique;Caudal block or Quadratus lumborum block .The method used is often chosen by which one the doctor has more experience using. The Investigator plans to find out if one of the methods is more effective and/or safer than the other method.

The results of this study will help learn how to best control pain in children having surgery low abdominal surgery.

DETAILED DESCRIPTION:
Children aged 1-9 years undergoing lower abdominal surgeries would be recruited in this randomized study.

Children would be monitored by electrocardiogram, pulse oximeter and non-invasive blood pressure.

After preoxygenation for three minutes, anesthesia would be induced with 8% sevoflurane inhalation in 50% oxygen and % 50 air ; 1ug/kg fentanyl and 3 mg/kg propofol is administered intravenously. Then laryngeal mask is inserted when conditions are satisfactory (jaw relaxed, lash reflex disappeared, no coughing, gagging, swallowing).After ethical committee approval, informed written consent will be obtained from all patients.

Consenting patients scheduled to have unilaterally low abdominal surgery(inguinal hernia,hydrocele,undescended testicles surgery will be randomised to unilateral Quadratus lumborum block or caudal block at the begin of surgery.

All patients heart rate,MAP and Oxygen saturation record intraoperatively. All patients will receive paracetamol if requirement for postoperative analgesia.All patient will transfer from PACU to day-surgery unit (DSU) if they achieved Modified Aldrete Score of ten.

All patients will be assessed postoperatively by a blinded investigator: in the postanesthesia care unit and at 30 min 1,2, 4, 6, 12, 24, hour postoperatively.FLACC and Modified Children's Hospital of Eastern Ontario Pain Scale (CHEOPS) score will be used.

ELIGIBILITY:
Inclusion Criteria:

1. Age 1-9
2. ASA physical status I-II
3. Undergoing unilateral low abdominal surgery

Exclusion Criteria:

1. History of developmental delay or mental retardation, which will make observational pain intensity assessment difficult
2. Parent refusal
3. History of allergic reactions to local anesthetics
4. Rash or infection at the injection site
5. Anatomical abnormality
6. Bleeding diatheses
7. Coagulopathy,
8. History of diseases

   1. renal
   2. hepatic
   3. cardiac
   4. upper or lower airway
   5. neurological

Ages: 1 Year to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Use of analgesic consumption | 24 hour
  paracetamol

SECONDARY OUTCOMES:
Flacc score( face, legs, activity, cry, consolability) | 1,2,4,6,12,24 hou
  By investigators until hospital discharge, then through telephone interview with parents after that
Parent satisfaction scores | 24 hour
  By investigators until hospital discharge, then through telephone interview with parents after that
Time to first use of analgesic | 24 hour
  By investigators until hospital discharge, then through telephone interview with parents after that

CONTACTS AND LOCATIONS:
Overall Officials: Gözen Öksüz, M.D., Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- KahramanmarasSIU, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Oksuz G, Bilal B, Gurkan Y, Urfalioglu A, Arslan M, Gisi G, Oksuz H. Quadratus Lumborum Block Versus Transversus Abdominis Plane Block in Children Undergoing Low Abdominal Surgery: A Randomized Controlled Trial. Reg Anesth Pain Med. 2017 Sep/Oct;42(5):674-679. doi: 10.1097/AAP.0000000000000645. PMID 28759502
- [Derived] Oksuz G, Arslan M, Urfalioglu A, Guler AG, Teksen S, Bilal B, Oksuz H. Comparison of quadratus lumborum block and caudal block for postoperative analgesia in pediatric patients undergoing inguinal hernia repair and orchiopexy surgeries: a randomized controlled trial. Reg Anesth Pain Med. 2020 Mar;45(3):187-191. doi: 10.1136/rapm-2019-101027. Epub 2020 Jan 5. PMID 31907294